CLINICAL TRIAL: NCT06059729
Title: Effect of Al-Lisaan Digital Application on Adult Stutters
Brief Title: Effects of Al-Lisaan Urdu Digital Software for Self-Assessment and Treatment of Adult Stutters
Acronym: Al-Lisaan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 27231-Hafsa Noreen
Record Dates: First submitted 2023-09-22; First posted 2023-09-29 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Stuttering, Adult
MeSH Terms: conditions — Stuttering

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Al-Lisaan digital application will be given to participants for self assessment and management
  Interventions: Device: Al-Lisaan
- Controlled group (Other): Home plan will be given
  Interventions: Device: Al-Lisaan

INTERVENTIONS:
Device: Al-Lisaan — Al-Lisaan is a digital application for the self assessment and management of adult stutters.

SUMMARY:
The study plans to find the efficacy of a digital application/software, Al-lisan that adult stutters can be used for assessment and management of their stuttering. The Software has been developed with the help of a software engineer. After the current trends employed by Speech language pathologists explored through qualitative study design, the manual which is under development process through a focused group in which assessment and treatment options of the software were finalized. The next step will include the reliability and validity of the software for assessment and management of adult stutters followed by finding the efficacy of the software. As this Application will be in Urdu language it will assist less literate and those living in peripheries to assess or provide self-treatment options to the persons who stutter. It will allow adults for self-assessment and treatment options in Urdu language.

DETAILED DESCRIPTION:
The term stuttering refers to the dis-fluent pattern of speech. In adult stuttering it's a learned pattern of dis-fluent production that may become the part of their speech permanently. It affects 1% of the worldwide population. There are many therapeutic techniques to treat the stuttering in adults. Self-help therapy is common to use. Besides the personalized treatment of self-help therapy by adult stutters, there are many digital applications available and used by many adult stutters worldwide. Few are StammerApp, Stamurai and SMAAT. The objective of the study is to develop a digital application/software that adult stutters can be used for assessment and management of their stuttering. This study being a part of PhD project, started in March 2020 and until now, the current trends employed by Speech language pathologists have been explored through qualitative study design. The manual was developed through a focused group in which assessment and treatment options of the software were finalized. The Software has been developed with the help of a software engineer. The objective of this study is to find the effects of Al-lisan Urdu Digital Software for Self-Assessment and Treatment of Adult Stutters. For this step we are applying for the grant. As this Application will be in Urdu language it will assist less literate and those living in peripheries to assess or provide self-treatment options to the persons who stutter. It will allow adults for self-assessment and treatment options in Urdu language.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria will be Stutters who are above the age of 19 and who have not taken regular therapy from last one year

Exclusion Criteria:

Adults with neurogenic stuttering or any other organic cause will be excluded

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Stutter Severity Index | six weeks
  Stutter's severity will be measured Pre and Post experimental study.

SECONDARY OUTCOMES:
Stuttering Severity Index | six weeks
  Stutter's severity will be measured Pre and Post experimental study.

CONTACTS AND LOCATIONS:
Overall Officials: hafsa Noreen, PhD*, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Hafsa Noreen, Lahore, Punjab Province
  - Rex Medical Center, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No